CLINICAL TRIAL: NCT00026624
Title: A Phase I/II Study to Evaluate the Safety and Immunogenicity of the Subcutaneous Administration of ALVAC-HIV vCP1452 Infected Autologous Dendritic Cells Versus the Subcutaneous Administration of ALVAC-HIV vCP1452 To HIV-Infected Subjects
Brief Title: Safety/Immunogenicity of Immunizations of ALVAC-DC-SC vs ALVAC-SC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A5130; AACTG A5130; 10080 (Registry Identifier: DAIDS ES Registry Number); ACTG A5130
Record Dates: First submitted 2001-11-12; First posted 2001-11-13 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; Injections, Subcutaneous; HIV-1; AIDS Vaccines; Dendritic Cells; Adoptive Transfer; Keyhole-Limpet Hemocyanin; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections | interventions — keyhole-limpet hemocyanin

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)
Drug: Keyhole-Limpet Hemocyanin

SUMMARY:
The purpose of this study is to determine how safe it is to give patients a shot that has a mixture of a vaccine and dendritic cells (DCs), a special kind of immune cell, and how safe it is to give a shot of the vaccine alone.

Current HIV vaccines have not been strong enough to give good immune responses. Research has shown that the immune response to a vaccine delivered by DCs is greater than the response without DC delivery. A5130 is a study that seeks to give good delivery of the vaccine to important immune cells of the body.

DETAILED DESCRIPTION:
Cytotoxic T-cell lymphocyte (CTL) responses are important in viral destruction and thereby in the protective immune response to viral infection. Current HIV vaccines do not consistently elicit strong CTL responses. The limited immune response of current HIV vaccines could be attributed, in addition to other causes, to failure of the vaccine to reach the appropriate cells to initiate a robust immune response. DCs particularly are effective in stimulating primary T-cell-dependent immunity. Antigen-bearing DCs are used as adjuvants for active immunotherapy in humans, particularly to increase host resistance to tumors and certain viral infections. A5130 is an exploratory, proof-of-concept study that seeks to ensure adequate delivery of the vaccine to important antigen-presenting cells.

Patients are randomized into 1 of 2 vaccination groups at entry. Group A: Patients receive an SC vaccination with DCs infected with ALVAC-HIV vCP1452. DC exposure to KLH occurs at Weeks 3 and 7. Leukopheresis occurs at entry.

Group B: Patients receive an SC vaccination with ALVAC-HIV vCP1452 without DCs. KLH injections are administered at Weeks 3 and 7.

Patients in both groups receive their vaccinations at Weeks 3, 7, and 15. This study consists of 4 steps but not all patients necessarily qualify to enter Step II, Step III, or Step IV.

Step I: vaccination phase. Step II: withdrawal of potent ART. Step III: optional discontinuation of ART. Step IV: reinitiation of ART. [AS PER AMENDMENT 04/10/02: Step V: follow-up period off potent ART.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-infected.
* Took 3 or more anti-HIV drugs for 3 or more months before study entry.
* Have a viral load of 400 copies/ml or less for a period of 3 months before study start and within 30 days before study start.
* Have a CD4 count of 400 cells/mm3 or more for a period of 3 months before study start and within 30 days before study start.
* Have a CD4 count of 400 cells/mm3 or more at study screening.
* Have a viral load of 50 copies/ml or less at study screening.
* Are at least 18 years old.
* Agree not to become pregnant or to impregnate during the study and for 12 weeks after the study, if able to have children.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have a short-term but intense infection or serious illness within 14 days before study start and have not completed therapy or are not clinically stable on therapy.
* Have viral load values greater than 400 copies/ml within 3 months before study start.
* Have CD4 counts less than 400 cells/mm3 within 3 months before study start.
* Have close contact with canaries through work (e.g., breeding farms, bird shops). Does not apply to pet canaries.
* Are allergic to eggs or neomycin. Have a history of serious allergic reactions including allergy-induced asthma.
* Are sensitive or allergic to study drugs.
* Use drugs or alcohol in a way that would interfere with the patients' ability to follow the study requirements.
* Have become HIV-positive within 1 year before study start.
* Are pregnant or breast-feeding.
* Have had lymph node irradiation.
* Have had any HIV vaccine.
* Have used hydroxyurea within 45 days of study start.
* Have received drugs that affect the immune system, such as corticosteriods, within 30 days before study start.
* Are allergic to shellfish. (This study has been changed to make shellfish allergy an exclusion criterion and to remove abacavir use as an exclusion criterion.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jacobson, Study Chair
Locations (2):
- United States (2):
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Med. Ctr., ACTU, New York, New York

REFERENCES:
- [Derived] Gandhi RT, O'Neill D, Bosch RJ, Chan ES, Bucy RP, Shopis J, Baglyos L, Adams E, Fox L, Purdue L, Marshak A, Flynn T, Masih R, Schock B, Mildvan D, Schlesinger SJ, Marovich MA, Bhardwaj N, Jacobson JM; AIDS Clinical Trials Group A5130 team. A randomized therapeutic vaccine trial of canarypox-HIV-pulsed dendritic cells vs. canarypox-HIV alone in HIV-1-infected patients on antiretroviral therapy. Vaccine. 2009 Oct 9;27(43):6088-94. doi: 10.1016/j.vaccine.2009.05.016. Epub 2009 May 29. PMID 19450647